CLINICAL TRIAL: NCT01748201
Title: Viscosupplementation in Patients With Hemophilic Arthropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0199/11
Record Dates: First submitted 2012-12-06; First posted 2012-12-12 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Osteoarthritis; Hemarthrosis; Hemophilia A; Hemophilia B
Keywords: Osteoarthritis; Hemarthrosis; Hemophilia A; Hemophilia B; Viscosupplementation
MeSH Terms: conditions — Osteoarthritis; Hemarthrosis; Hemophilia A; Hemophilia B | interventions — Viscosupplementation; Injections, Intra-Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Joint lavage and viscosupplementation (Experimental): The joint will be washed until obtaining translucent liquid and not hemorrhagic. Then it will receive an intra-articular injection of 6ml of hyaluronic acid (Synvisc One), 1ml of triamcinolone and 2 ml of ropivacaine.
  Interventions: Procedure: Joint lavage and viscosupplementation

INTERVENTIONS:
Procedure: Joint lavage and viscosupplementation — The joint will be washed until obtaining translucent liquid and not hemorrhagic. Then it will receive an intra-articular injection of 6ml of hyaluronic acid (Synvisc One), 1ml of triamcinolone and 2 ml of ropivacaine.
  Other Names: intra-articular injection

SUMMARY:
Hemophilia is a recessive X chromosome linked genetic disorder of blood coagulation that affects about one in every ten thousand people. Hemarthrosis, which you can begin in childhood, promptly leads to degenerative changes of the articular cartilage which culminate in deformity and degenerative changes early, known as hemophilic arthropathy, which is the most common complication of hemophilia. Aside administration of clotting factor, treatment should address the degenerative changes already present in patients joints. Our objective is to evaluate the effectiveness of articular washing followed by infiltration with corticosteroids and hylan G-F 20, followed by a program of home exercises and/or academy as the previous level of hemophilia patients, in relation to pain relief, and improved function and quality of life.

DETAILED DESCRIPTION:
Hemophilia is a recessive X chromosome linked genetic disorder of blood coagulation that affects about one in every ten thousand people. There are two main types of hemophilia. Hemophilia A or classical hemophilia corresponds to 80% of the cases, and is caused by a deficiency or change of factor VIII. Hemophilia B is caused by deficiency or amendment of factor IX, and represents about 20%. Patients with hemophilia type A or B have the same clinical presentation. Cases with moderate or severe hemophilia exhibit a tendency to spontaneous bleeding or after minimal trauma, being the joints the most frequent sites of hemorrhage. The joints most commonly affected are the knees, followed by the elbows, ankles, shoulders and hips. Hemarthrosis, which you can begin in childhood, promptly leads to degenerative changes of the articular cartilage which culminate in deformity and degenerative changes early, known as hemophilic arthropathy, which is the most common complication of hemophilia. The hemophilic arthropathy is highly debilitating and consumes a large amount of resources for the treatment of hemophilic patients. Currently, by the adequate administration of the clotting factor, the hemophilic patient has a life expectancy of next to normal. Therefore other forms of treatment must be researched; they can be palliative or modifiers of the natural history of disease, to try to postpone the need for arthroplasty . Our objective is to evaluate the effectiveness of treatment, consisting of articular washing followed by infiltration with corticosteroids and hylan G-F 20, followed by a program of home exercises and/or academy as the previous level of hemophilia patients, in relation to pain relief, and improved function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patients with hemophilia A or B;
* symptomatic arthropathy;

Exclusion Criteria:

* inadequate follow-up;
* Bleeding elsewhere as to not allow for functional evaluation;
* complications of Arthrocentesis (infection).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
WOMAC | 12 months
  Evaluation of patient's symptoms using Western Ontario and McMaster Universities osteoarthritis index (WOMAC
VAS | 12 months
  Visual analogic scale for pain assessment
Lequesne | 12 months
  Evaluation of patient's symptoms using Lequesne questionaire

SECONDARY OUTCOMES:
SF-36 | 12 months
  Evaluation of patient's quality of life using the quality of life's questionaire (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia U Rezende, Phd, Principal Investigator — FMUSP
Locations (1):
- Instituto de Ortopedia e Traumatologia HC-FMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Brazilian Orthopaedics Association — http://sbot.org.br
- See also: Orthopaedics and Traumatology Institute website — http://www.iothcfmusp.com.br